CLINICAL TRIAL: NCT04633525
Title: A Prospective Study to Define Optimum Cup Orientation in Hip Arthroplasty Accounting for the Individual's Anatomy and Movement Patterns
Brief Title: Defining Optimum Cup Orientation for Hip Replacements Taking Into Account the Individual's Anatomy and Movement Patterns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2251
Record Dates: First submitted 2020-08-11; First posted 2020-11-18 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Hip Arthritis; Hip Osteoarthritis
Keywords: Hip Replacement; Hip Arthroplasty; Arthritis; Osteoarthritis; Hip dislocation
MeSH Terms: conditions — Osteoarthritis, Hip; Arthritis; Osteoarthritis; Hip Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Optimum Cup Orientation (Experimental)
  Interventions: Procedure: Optimum Cup Orientation

INTERVENTIONS:
Procedure: Optimum Cup Orientation — Participants will have X-rays taken before surgery to determine the target optimal zone for orientation of the cup implant, using EBRA software. The surgeon may or may not implant in this target zone, depending on what they believe is in the patient's best interest. X-rays will be taken at 12 months after surgery to determine if they target cup orientation was achieved.

SUMMARY:
The purpose of this study is to investigate and determine the optimal zone for implanting the cup component (the ball that sits in the joint socket) in a total hip replacement. Enrolled participants will have a series of X-rays analyzed before surgery to identify their individual optimal zone or cup orientation. This information will be provided to the operating surgeon, who may use this information to influence the placement of the cup implant. Follow-up X-rays taken after surgery will determine if the cup is within the suggested optimal zone. Questionnaires will be completed before and after surgery, and data on complications or issues with the surgery (including incidents of dislocation) will be collected after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Signed up for primary total hip arthroplasty procedures at the General Campus at The Ottawa Hospital.

Exclusion Criteria:

* Unwilling or unable to complete study requirements (either X-rays or questionnaires)
* Unwilling or unable to sign the informed consent form

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-11-18 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Cup Orientation | 12 months after surgery
  The degree of cup inclination and anteversion as shown on X-rays

SECONDARY OUTCOMES:
Change in Patient Reported Function | 12 months
  Assess the change in function using the Oxford Hip Score. Total scores range from 0-48. The higher the score, the better the outcome.
Change in Patient Reported Pain | 12 months
  Assess the change in pain using the Oxford Hip Score. Total scores range from 0-48. The higher the score, the better the outcome.
Change in Patient Reported Health | 12 months
  Assess the change in general health using the EQ-5D-5L
Change in Patient Reported Health | 12 months
  Assess the change in general health using the PROMIS-15
Incidence of Adverse Events | Up to 12 months after surgery
  Assess safety and post-operative complications by collecting information on adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: George Grammatopoulos, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada